## Athens Greece 15. 11. 2024

ClinicalTrials.gov ID: NCT05623228

Brief Title: The Effectiveness and Efficacy of the Combination of the Integrated

Psychological Therapy and Metacognitive Training. (ATHSCHIZ) (ATH22-24)

Official Title: The Effectiveness and Efficacy of the Combination of the

Integrated

Psychological Therapy and Metacognitive Training in Schizophrenia and

Treatment Resistant Schizophrenia. This is a Non-randomized Trial. The

Therapy Lasts 60 Sessions.

Dr. Stavroula Rakitzi

Clinical psychologist and cognitive behavioral psychotherapist

Private practice

ILISION 34

15771 Athens Greece

Tel: +306989766935

srakitzi@gmail.com

Links: URL: https://www.linkedin.com/

Description linkedin Stavroula Rakitzi

URL: http://orcid.org

Description orcid: 0000-0002-5231-6619

Psychiatrist and cognitive behavioral psychotherapist

Private practice

ILISION 34

15771 Athens Greece

Tel: +306932905259

polyxenigeorgila@gmail.com

Links: URL: https://www.linkedin.com/

Description linkedin Polyxeni Georgila

URL: http://orcid.org

Orcid:0000-0003-3137-506X

The aim of this study was to evaluate the effectiveness of the combination of Integrated psychological Therapy and the metacognitive training for psychosis. All the subprograms of IPT in 50 sessions and 10 sessions of MCT were offered in two biweekly one-hour sessions. 35 patients with schizophrenia took part in this study. Cognition, symptoms, functional outcome and recovery were assessed with a test battery before the therapy, after the therapy and in a follow-up after 6 months. General linear model and regression analysis were used. Significant effects were found in neurocognition, symptoms, functional outcomes and recovery. Effect sizes were also calculated. Significant effects were also found for the subgroup with treatment resistant schizophrenia in neurocognition, social cognition, symptoms, functional outcome and recovery. Effect sizes were also calculated. This study supports evidence for the effectiveness of the combination of IPT and MCT in Greece.

#### 1. Introduction

Schizophrenia presents a chronic mental health disorder with a high vulnerability and a huge emotional and social burden. Schizophrenia and especially treatment resistant

schizophrenia (TRS) needs evidence-based and recovery-oriented pharmacotherapy and cognitive behavioral psychotherapy and rehabilitation. Pharmacotherapy presents the main therapy for patients with schizophrenia (Huhn et al., 2019; Leucht et al., 2013; Taipale et al., 2018; Wagner et al., 2021). The Integrated Psychological Therapy (IPT) presents an efficacious evidencebased rehabilitation program for patients with schizophrenia (Roder et al., 2008, 2010, 2011, 2013). It is also translated in Greek (Roder, 2007). Our research group has implemented Integrated Psychological Therapy (IPT) the last years in Greece (Rakitzi et al., 2016, 2019, 2020, 2021). There are also other research groups in Greece that implemented IPT (Poulou, 2024). In other words, IPT is well known and established in Greece.

Metacognitive Training (MCT) for Psychosis presents also an efficacious and evidence-based therapy for people with schizophrenia and other psychotic disorders (Moritz et al., 2022; Penney et al., 2022; Veckenstedt & Scheunemann, 2023). MCT is implemented nowadays also in other mental health disorders, such as bipolar disorder and depression.MCT for psychosis is implemented for the first time in Greece in this research

project. This is also the first study, as far as it is known, in which IPT will be combined with MCT.IPT and MCT present two therapy programs which are used in our private practice systematically. The main hypothesis is: The combination of IPT and MCT is effective and

efficacious. The therapy shows improvement in cognition (neurocognition, social cognition), in psychopathology, in functional outcome and recovery.

#### 1. Material and methods

## 2.1. Compliance with ethical standards

The patients have given written informed consent for their participation in this research project prior to the inclusion of the study. Details which might disclose the identity of the patients were omitted. The authors follow the APA ethical standards.

The authorities in Greece does not prohibit the conducting of research protocols from scientists who treat patients in a private practice. There is no ethical commission which evaluates research projects from scientists in the private sector.

## 2.2. Study population

The outpatients with schizophrenia were recruited from Dr. P. Georgila psychiatrist and cognitive behavioral psychotherapist and Dr. S. Rakitzi clinical psychologist and cognitive behavioral psychotherapist from their own private practice. All participants were treated by both authors ambulant the last 15 years. All participants are treated monthly by Dr. P. Georgila and participated in individual cognitive behavioral psychotherapy of 30 sessions in the past by Dr. S. Rakitzi.

A motivational interview was conducted with all the patients from Dr. Georgila and Dr. Rakitzi to enhance their motivation for participating in a group cognitive behavioral psychotherapy and rehabilitation. The patients have given written informed consent for their participation in this research project, and they were not paid for their participation. A total of 35 patients with schizophrenia participated in this study.

The inclusion and exclusion criteria of the study were the following: inclusion criteria: patients with schizophrenia between 19-60 years old, an IQ over 80 and patients must be treated in an ambulant psychiatric treatment. Exclusion criteria: Relapse and hospitalization, substance abuse and diagnosis of other psychotic disorders.

Finally, pharmacotherapy was not changed from Dr. P. Georgila during the therapy, after the therapy and in the follow-up evaluation.

### 2.3. Study design

and were allocated to the therapy group. Afterwards, they were evaluated in post therapy after 60 sessions (T2) and at a follow up of 6 months after the end of the therapy (T3).

# 2.4. Therapists

Dr, P. Georgila and Dr. S. Rakitzi were the therapists. Dr. Georgila was the main therapist for the subprograms of IPT cognitive differentiation, social perception and verbal communication and Dr. S. Rakitzi the co-therapist. Dr. S. Rakitzi was the main therapist for the subprograms of IPT social skills and problem-solving and for the MCT for psychosis. Dr. P. Georgila was co-therapist. Both therapists are well trained by IPT and MCT.

#### 2.5. Intervention

IPT is a group therapy for patients with schizophrenia and contains 5 subprograms: Cognitive differentiation (neurocognition), social perception (social cognition), verbal communication, social skills and interpersonal problem-solving and presents an efficacious and evidence-based program for patients with schizophrenia (Roder et al., 2008, 2010). IPT was translated in Greek and was implemented with success from our research group (Rakitzi et al., 2016, 2019, 2020, Roder et al., 2007. IPT was implemented also from other research groups in Greece with very good results (Poulou et al., 2024). In other words, IPT is well known and established in Greece.

All 5 subprograms of IPT in 50 biweekly sessions of 1 hour were implemented in this study.

MCT presents an efficacious and evidence-based group rehabilitation program for many mental health disorders. 10 biweekly sessions of one hour of MCT for psychosis were implemented in this study after IPT. It is the first implementation of MCT in Greece.

The implementation of this therapy was conducted in 8 small groups: 1 (5 patients), 2(2 patients), 3(8 patients), 4(8 patients), 5(3 patients), 6(3 patients), 7(3 patients), 8(3 patients).

## 2.6. Measures

#### 2. 6. 1 WAIS

WAIS was implemented to all patients from Dr. S. Rakitzi for the evaluation of IQ before

the baseline assessment of this research project (Aster. 2006).

## 2. 6. 2. Cognition (proximal outcome)

Neurocognition (speed of processing, working memory, visual memory, reasoning and problem-solving) of MCCB were used. Working memory was evaluated with the Letter Number Span using the Greek translation (Gold et al., 1997; Nuechterlein & Green, 2006, Rakitzi, 2007a). The Greek verbal memory test was used to evaluate verbal memory-oral and written (Kosmidou, 2010). Social cognition (MSCEIT-emotional intelligence) of MCCB (Nuechterlein & Green, 2006) and social perception scale using the Greek translation were also used (Garcia et al., 2003; Rakitzi et al., 2007b; Ruiz et al., 2005). A blinded rater (Msc. Clinical psychology) has given the above tests before the therapy, after the therapy and in the follow-up of 6 months.

## 2.6.3. Psychopathology (proximal outcome)

Psychopathology was evaluated from PRYRAT (Haddock et al., 1999) and PANSS (Lykouras et al., 2005). A blinded rater (M. D.) has conducted the PSYRAT and PANSS before the therapy, after the therapy and in the follow-up after 6 months.

## 2.6.4. Functional outcome (proximal outcome)

Functional outcome was from WHODAS evaluated (Koumpouros et al., 2018; WHO, 2001). A blinded rater (Msc. Clinical psychology) has given the above tests before the therapy, after the therapy and in the follow-up of 6 months.

# 2.6.5. Recovery (proximal outcome)

Recovery was evaluated from the Greek version of RAS-DS (Hancock et al., 2019, 2023). RAS-DS is a reliable and valid scale (Hancock et al., 2015, 2019; Honey et al., 2023; Ramesh et al., 2024). A blinded rater (Msc. Clinical psychology) has given the above tests before the therapy, after the therapy and in the follow-up of 6 months.

### 2. 7. Statistical analysis

SPSS version 13 has been used for statistical analysis. A general linear model for repeated measures was chosen. A general linear model understands and quantifies the relationship between therapy and the proximal outcomes. A Bonferroni correction was made. Confounding variables were controlled. A regression analysis was conducted. A

regression analysis quantifies the strength between the variables (therapy and proximal outcomes) Effect sizes were also calculated. A statistical analysis (general linear model, effect sizes, regression analysis) was conducted for the 35 participants and afterward a second analysis was conducted (general linear model, effect sizes, regression analysis) focusing on the group of treatment resistant schizophrenia (Bortz & Döring, 2002; Cohen, 1988).

#### References

Aster, M., Neubauer, M., & Horn, R. (2006). Wechsler-Intelligenztest für Erwachsene WIE. Frankfurt: Harcourt Test Services

Bortz, J., & Döring, N. (2002). Forschungsmethoden und Evaluation für Human- und Sozialwissenschaftler. Berlin: Springer.

Cohen, J. (1988). Statistical Power Analyses for Behavioural Sciences. Erlbaum, Hillsdale, NJ.

Fuentes, I., Garcia, S., Ruiz, J.C., Soler, J., & Roder, V. (2007). Social perception scale in Schizophrenia. A pilot study. *International Journal of Psychology and Psychological therapy*, *7* (1), 1-12.

Garcia, S., Fuentes, I., Ruiz, J.C., Gallach, E., & Roder, V. (2003). Application of the IPT in a Spanish sample: evaluation of the "social Perception subprogram". International Journal of psychology and psychological therapy, 3(2), 299-310.

Haddock, G., McCarron, J., Tarrier, N., & Faragher E.B. (1999). Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). *Psychological Medicine*, *29(4)*, 879-889.

Hancock, N., Scanlan, J.N., Bundy, A.C., & Honey A. (2019). *Recovery Assessment Scale –Domains & Stages (RAS–DS) Manual- Version 3*. Sydney: University of

Sydney.

Hancock, N., the University of Sydney, Rakitzi, S. & Katoudi, S. (2023). *Recovery Assessment Scale-Domains & Stages (RAS-DS)*. The Greek version.

Hancock, N., Scanlan, J., Honey, A., Bundy, A., & O'Shea, K. (2015). Recovery Assessment Scale – Domains & Stages (RAS-DS): Its Feasibility and Outcome Measurement Capacity.

\*\*Australian\*\* and New Zealand Journal of Psychiatry, 49(7), 624633.http://dx.doi.org/10.1177/0004867414564084

Honey, A., Hancock, N., & Scanlan, J.N. (2023). Staff perceptions of factors affecting the use of RAS-DS to support collaborative mental health practice. *BMC Psychiatry*, *23*, 500 . https://doi.org/10.1186/s12888-023-04996-2.

Huhn, M., Nikolakopoulou, A., Schneider-Thoma, J., Krause, M., Samara, M., Peter, N., & Leucht S, et al. (2019). Comparative efficacy and tolerability of 32 oral antipsychotics for the acute treatment of adults with multi-episode schizophrenia: a systematic review and network meta-analysis. *Lancet*, *394*, 939-951. doi:10.1016/S0140-6736(19)31135-3

Kosmidou, M., & Vlahou, C. (2010). *Greek verbal memory test.* Athens: Parisianos.

Koumpouros, Y., Papageorgiou, E., Sakellari, E. et al. (2018). Adaptation and psychometric properties' evaluation of the Greek version of WHODAS 2.0. Pilot application in Greek elderly population. *Health Services and Outcomes Research Methodology*, *18*(1), 63-74. https://doi.org/10.1007/s10742-017-0176-x.

Leucht, S., Cipriani, A., Spineli, L., Mavridis, D., Őrey, D., Richter, F., Davis, J.M. et al. (2013). Comparative efficacy and tolerability of 15 antipsychotic drugs in schizophrenia: a multiple-treatments meta-analysis. *Lancet*, *382*(9896), 951-962.

# https://doi.org/10.1016/S0140-6736(13)60733-3.

Lykouras, L., Botsis, A., & Oulis, P. (2005). *Greek version of PANSS*. Athens: Scientific publications.

Moritz, S., Menon, M., Balzan, R., & Woodward, T.S. (2022). Metacognitive training for psychosis (MCT): past, present and future. European Archives of Psychiatry and Clinical Neurosciences. https://doi.org/10.1007/s00406-022-01394-9.

Mueller, D.H., Schmidt, S.J., & Roder, V. (2013). Integrated Psychological Therapy. Effectiveness in schizophrenia inpatient settings related to patients age. *American Journal of Geriatric Psychiatry, 21(3),* 231-241. http://dx.doi.org.10.1016/j.jagp.2012.12.011.

Nuecterlein, K. H., & Green, M. F. (2006). *MCCB. MATRICS Consensus Cognitive Battery*. LA: MATRICS Assessment Inc.

Penney, D., Sauvé, G., Mendelson, D., Thibaudeau, E., Moritz, S., & Lepage, M. (2022). Immediate and sustained outcomes and moderators associated with metacognitive training for psychosis. A systematic Review and Meta-analysis. *JAMA Psychiatry* doi:10.1001/jamapsychiatry.2022.0277.

Poulou, A., Anagnostopolos, Fotios., Vatakis, A., Mellon, R. C., & Mueller, D. R. (2024). The implementation and effectiveness of Integrated Psychological Therapy (IPT) in chronic middle-aged inpatients with schizophrenia. Schizophrenia Research: Cognition 39 (2025) 100330. <a href="https://doi.org/10.1016/j.scog.2024.100330">https://doi.org/10.1016/j.scog.2024.100330</a>.

Rakitzi, S., Georgila, P., Efthimiou, K., & Müller, D.R. (2016). Efficacy and feasibility of the Integrated Psychological Therapy for outpatients with schizophrenia in Greece: Final results of a RCT. *Psychiatry Research*, *242*, 137-143. http://dx.doi.org/10.1016/j.psychres.2016.05.039.

Rakitzi, S., & Georgila, P. (2019). Integrated Psychological Therapy and Treatment Resistant Schizophrenia: Initial Findings. Psychiatry, 82(4), 354-367.

Rakitzi, S., Georgila, P., & Becker-Woitag, A.P. (2021). The Recovery Process for Individuals with schizophrenia in the context of evidence-based psychotherapy and rehabilitation. *European Psychologist*, *26*(2), 96-111. <a href="https://doi.org/10.1027/1016-9040/a000400">https://doi.org/10.1027/1016-9040/a000400</a>.

Rakitzi S. (2020). Grundlagen evidenzbasierter Rehabilitation von Schizophrenieerkrankten. Basics of evidence-based Rehabilitation in individuals with schizophrenia. Doctoral thesis. Universität Koblenz-Landau, Campus Landau, Universitätsbibliothek.

Rakitzi S. (2023). Clinical Psychology and Cognitive Behavioral Psychotherapy.

Recovery in Mental Health. Cham, Switzerland: Springer.

Rakitzi, S., & Georgila, P. (2024). *Treatment resistant schizophrenia. Evidence-based pharmacotherapy, cognitive behavioral psychotherapy and rehabilitation.* Cham: Springer Nature.

Rakitzi, S. (2007a). The Letter Number Span in Greek. Translation. Unpublished.

Rakitzi, S. (2007b). The Social Perception Scale in Greek. Unpublished.

Ramesh, S., Scanlan, J.N., Honey, A., & Hancock, N. (2024). Feasibility of Recovery Assessment Scale-Domains and stages (RAS-DS) for every day mental health practice. *Frontiers in Psychiatry*, *15*, 1256092. doi: 10.3389/fpsyt.2024.1256092

Roder, V., Brenner, H.D., Kienzle, N., & Efthimiou, K. (2007). *The GREEK manual of Integrated Psychological Therapy. (I. P. T.)*. Athens: Scientific Publications.

Roder, V., Brenner, H.D., Kienzle, N., 2008. Integriertes Psychologisches Therapieprogramm bei schizophren Erkrankten. IPT. Beltz, Weinheim.

Roder, V., Mueller, D.R., Brenner, H.D., & Spaulding, W. (2010). *Integrated Psychological* 

Therapy (IPT) for the Treatment of Neurocognition, Social Cognition and Social Competency in Schizophrenia Patients. Seattle: Hogrefe & Huber.

Roder, V., Mueller, D.R., & Schmidt, S.J. (2011). Effectiveness of Integrated Psychological

Therapy (IPT) for schizophrenia patients. *Schizophrenia Bulletin, 37 (Suppl. 2),* S71-S79.

Taipale, H., Mehtälä, J., Tanskanen, A., & Tiihonen J. (2018). Comparative effectiveness of antipsychotics drugs for rehospitalization in schizophrenia. A Nationwide study with 20 year follow up. *Schizophrenia Bulletin, 44(6),* 1381-1387.doi: 10.1093/schbul/sbx176.

Veckenstedt, R., Scheunemann, J. (2023). Metakognitives training für Patientinnen mit Psychose in Gruppen- und Einzelsetting. *Psychotherapeut*, *3*, 255-260.

Wagner, E., Siafis, S., Fernando, P., Falkai, P., Honer, W.G., Röh, A., Siskind, D., Leucht, S., & Hasan, A. (2021). Efficacy and safety of clozapine in psychotic disorders.